CLINICAL TRIAL: NCT02848196
Title: A Phase II Trial of Image-guided Stereotactic Body Radiation Therapy (SBRT) for Adrenal Gland Metastasis in Oligometastatic Patients
Brief Title: An Image-guided SBRT for Adrenal Gland Metastasis in Oligometastatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1580
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Adrenal Gland Metastases
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic body radiation therapy (Experimental): Oligometastatic patients with adrenal gland metastases are treated with high dose of Stereotactic Body Radiation Therapy delivered with VMAT/Rapid Arc technique.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — The schedule will be 3 fractions of 15 Gy up to a total dose of 45 Gy delivered every day with VMAT and Flattening filter-free (FFF) beams. Image-guided systems, including CBCT, will be used for all patients.

SUMMARY:
The study is designed to to assess the efficacy of ablative SBRT delivered with VMAT technique in oligometastatic patients affected by adrenal gland metastases.

DETAILED DESCRIPTION:
This is a phase II, single arm, trial for testing efficacy of ablative high hypofractionated dose delivered with VMAT technique in oligometastatic patients with adrenal gland metastases. The potential advantages of this approach include the possibility to lead an increased local control in irradiated adrenal gland metastases. Other purpose of this study is to assess acute and late toxicity in terms of maintenance of endocrine mechanisms of hormonal production.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years.
* WHO performance status ≤ 1 (ECOG - KPS).
* Histologically-proven of primary cancer disease
* Metastases at adrenal gland radiologically proven
* Written informed consent

Exclusion Criteria:

* Prior radiation to the interested adrenal gland.
* Patients allergic to contrast used in CT scans or who cannot be premedicated for the use of contrast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Control of local disease | 5 years
  Evaluation of proportion of patients free from progression from starting radiotherapy according to CTCAE v4.03

SECONDARY OUTCOMES:
Incidence of acute and late complications | 5 years
  Evaluation of early and late post treatment complications
Endocrine mechanisms of hormonal production | 5 years
  Assessment acute and late toxicity in terms of maintenance of endocrine mechanisms of hormonal production according to CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Franzese, MD, Principal Investigator — Humanitas Cancer Center
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No